CLINICAL TRIAL: NCT03100500
Title: A Multicenter, Open-label, Single Arm, 52-week Treatment Study to Assess the Safety of QMF149 in Japanese Patients With Asthma
Brief Title: A Long-term Safety Study of QMF149 in Japanese Participants With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQVM149B1305
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Asthma
Keywords: QVM149,; Asthma,; Japanese,; Allergic asthma,; Allergy triggered asthma,; Reactive asthma,; Asthma attack,; Difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea | interventions — QMF149

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QMF149 (Experimental): All eligible patients take QMF149 150/320 μg once daily over 52 weeks.
  Interventions: Drug: QMF149

INTERVENTIONS:
Drug: QMF149 — QMF149 150/320 μg once daily, delivered as powder in hard capsules via Concept1 inhaler

SUMMARY:
The purpose of this study was to provide long term safety data of QMF149 in Japanese participants with inadequately controlled asthma for the registration of QMF149 in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female adult patient ≥ 18 years old.
* Patients with a diagnosis of persistent asthma for a period of at least 1 year prior to Visit 1.
* Patients who have used medium or high dose inhaled corticosteroids (ICS) plus at least 1 controller for asthma for at least 3 months and at stable dose and regimen for at least 4 weeks prior to Visit 1.
* Patients must have Asthma Control Questionnaire-7 (ACQ-7) score ≥ 1.5 at Visits 2 and qualify for treatment with high dose ICS/long-acting β2 agonist (LABA).
* Pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) of ≥ 50% and ≤ 85% of the predicted normal value for the patient after withholding bronchodilators at Visit 2.
* Repeating is allowed once only. Repeating of percentage predicted FEV1 should be done in an ad-hoc visit to be scheduled on a date that would provide sufficient time to receive confirmation from the spirometry data central reviewer of the validity of the assessment before Visit 99.
* Patients must demonstrate reversibility defined as an increase in FEV1 of ≥ 12% and 200 mL within 15 to 30 minutes after administration of 400 µg of salbutamol at Visit 2. Spacer devices are permitted during reversibility testing only. The Investigator or delegate may decide whether or not to use a spacer for the reversibility testing.

  * If reversibility is not proven at Visit 2, patients may be permitted to enter the study with historical evidence of reversibility that was performed within 5 years prior to Visit 1.
  * Alternatively, patients may be permitted to enter the study with a historical positive bronchoprovocation test (defined as a provoked fall in FEV1 of 20% by bronchoconstriction agent e.g., methacholine, histamine) or equivalent test (e.g., astography) that was performed within 5 years prior to Visit 1.
  * Where patient is assessed as eligible based on historical evidence, a copy of the original printed report must be available as source documentation.
  * If reversibility is not proven at Visit 2 and historical data is not available, reversibility should be repeated once in an ad-hoc visit scheduled as close as possible from the first attempt (but not on the same day).
  * If reversibility is not demonstrated at Visit 2 (or after repeated assessment at ad-hoc visit) and historical evidence of reversibility/bronchoprovocation/astography is not available, patients must be screen failed.

Exclusion Criteria:

* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of Visit 1.
* Patients who have ever required intubation for a severe asthma attack/exacerbation.
* Patients who have a clinical condition which is likely to be worsened by ICS administration (e.g. glaucoma, cataract and fragility fractures) who are according to investigator's medical judgment at risk participating in the study.
* Patients who have had a respiratory tract infection or asthma worsening as determined by investigator within 4 weeks prior to Visit 1 or between Visit 1 and Visit 99. Patients may be re-screened 4 weeks after recovery from their respiratory tract infection or asthma worsening.
* Patients with a history of chronic lung diseases other than asthma, including (but not limited to) chronic obstructive pulmonary disease, sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Patients with severe narcolepsy and/or insomnia.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential unless they are using highly effective methods of contraception during dosing and for 30 days after stopping of investigational medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Japan (13):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Chitose, Hokkaido
  - Novartis Investigative Site, Kitahiroshima, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Chino, Nagano
  - Novartis Investigative Site, Higashiosaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- QMF-149 150/320 μg: QMF-149 150/320 μg delivered as powder in hard capsules, once daily via Concept1 inhaler.
Period: Overall Study
Arm/Group | QMF-149 150/320 μg
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Set consisted of all participants who received at least one dose of study medication during this study.
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  East Asian | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE is any adverse event that started on or after the time of the first inhalation of study drug but not later than 7 days (30 days in the case of a SAE) after the last administration. A SAE is described as any adverse event that leads to death, is life-threatening, results in persistent or significant disability/incapacity, causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event which is medically significant.
Time Frame: Up to 52 weeks
Population: Safety Set consisted of all participants who received at least one dose of study medication during this study.
Measure: Count of Participants; unit: Participants
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
Participants
  TEAEs | 40
  SAEs | 0

2. Secondary Outcome: Change From Baseline of Pre-Dose Forced Expiratory Volume in 1 Second (FEV1) Measured After 26 And 52 Weeks Treatment
Description: The pre-dose FEV1 was defined as the mean of the pre-dose 45 and 15 min FEV1 values prior to evening dose. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. A positive change from baseline in FEV1 indicates improvement in lung function.
Time Frame: Baseline, Weeks 26 and 52
Population: Full Analysis Set (FAS) consisted of all participants who entered the treatment epoch of this study and received at least one dose of study medication during this study. Participants with a value at both baseline and the respective day are included.
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
liters (L)
  Baseline | 2.1565 (0.58074)
  Change at Week 26: number analyzed (Participants) | 49
  Change at Week 26 | 0.2417 (0.26361)
  Change at Week 52: number analyzed (Participants) | 48
  Change at Week 52 | 0.1827 (0.26627)

3. Secondary Outcome: Change From Baseline of Morning and Evening Peak Expiratory Flow (PEF) During 52 Weeks Treatment
Description: PEF is the greatest airflow rate achieved during forced exhalation with lungs fully inflated. PEF was analyzed separately in the morning and evening using an electronic Peak Flow Meter (ePEF). A positive change from baseline in PEF indicates improvement in lung function.
Time Frame: Baseline up to Week 52
Population: FAS consisted of all participants who entered the treatment epoch of this study and received at least one dose of study medication during this study. Participants with a value at both baseline and the respective post baseline month are included.
Measure: Mean (Standard Deviation); unit: liters/minute (L/min)
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
liters/minute (L/min)
  Baseline, Morning PEF | 342.88 (94.656)
  Change through Weeks 1-52, Morning PEF | 15.49 (49.089)
  Baseline, Evening PEF | 352.65 (92.624)
  Change through Weeks 1-52, Evening PEF | 9.34 (42.685)

4. Secondary Outcome: Change From Baseline of Asthma Control Questionnaire (ACQ-7) After 26 And 52 Weeks Treatment
Description: The ACQ-7 is a seven-item disease-specific instrument developed and validated to assess asthma control in participants. It consists of five items to assess symptoms and activity limitations, one question to assess rescue medication use, and one question to assess airway caliber (FEV1% predicted). All seven items are scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating poor control. The questions are equally weighted and the total score is the mean of the seven items. The first 6 questions of the ACQ-7 were completed by the participant while the last question (question 7) was completed by the study investigator using data from the Master Scope spirometer. A negative change from baseline indicates improvement in lung function.
Time Frame: Baseline, Weeks 26 and 52
Population: FAS consisted of all participants who entered the treatment epoch of this study and received at least one dose of study medication during this study. Participants with a value at both baseline and the respective day are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
score on a scale
  Baseline | 1.983 (0.5381)
  Change at Week 26: number analyzed (Participants) | 50
  Change at Week 26 | -0.689 (0.6268)
  Change at Week 52: number analyzed (Participants) | 48
  Change at Week 52 | -0.830 (0.6852)

5. Secondary Outcome: Responder Rate of Participants Achieving the Minimal Important Difference (MID) of ACQ-7 ≥ 0.5 After 26 And 52 Weeks Treatment
Description: The ACQ-7 is a seven-item disease-specific instrument developed and validated to assess asthma control in participants. It consists of five items to assess symptoms and activity limitations, one question to assess rescue medication use, and one question to assess airway caliber (FEV1% predicted). All seven items are scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating poor control. The questions are equally weighted and the total score is the mean of the seven items. The first 6 questions of the ACQ-7 were completed by the participant while the last question (question 7) was completed by the study investigator using data from the Master Scope spirometer. The proportion of participants who achieved an improvement of at least 0.5 in ACQ-7 (i.e. decrease of ACQ-7 score of at least 0.5 from baseline) at post-baseline visits were analyzed.
Time Frame: Weeks 26 and 52
Population: FAS consisted of all participants who entered the treatment epoch of this study and received at least one dose of study medication during this study. Number analyzed indicates the number of participants with data available for analysis at Weeks 26 and 52.
Measure: Number; unit: percentage of participants
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
percentage of participants
  Week 26: number analyzed (Participants) | 50
  Week 26 | 66.0
  Week 52: number analyzed (Participants) | 48
  Week 52 | 72.9

6. Secondary Outcome: Change From Baseline of Rescue Medication Use During 52 Weeks Treatment
Description: Based on the electronic-diary data, the total number of puffs of rescue medication per day over the 52 weeks were calculated and divided by the total number of days to derive the mean daily number of puffs of rescue medication taken for the participant.
Time Frame: Baseline up to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: puffs/day
Arm/Group | QMF-149 150/320 μg
Number analyzed (Participants) | 51
puffs/day
  Baseline | 0.56 (1.382)
  Change through Weeks 1-52 | -0.18 (0.499)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: Safety Set consisted of all participants who received at least one dose of study medication during this study.
Groups:
- QMF149 150/320 µg: QMF-149 150/320 μg delivered as powder in hard capsules, once daily via Concept1 inhaler.
Arm/Group | QMF149 150/320 µg
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 37/51
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 150/320 µg (N=51)
Gastritis (Gastrointestinal disorders) | 2
Bronchitis (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 15
Otitis media (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 3
Electrocardiogram QT prolonged (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 28
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03100500/SAP_000.pdf
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03100500/Prot_001.pdf